CLINICAL TRIAL: NCT04247581
Title: ECG App Algorithms Clinical Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apple Inc. (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 013
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Results first posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Atrial Fibrillation
Keywords: Cardiovascular diseases; Heart Diseases; Arrhythmia; Cardiac
MeSH Terms: conditions — Atrial Fibrillation; Cardiovascular Diseases; Heart Diseases; Arrhythmias, Cardiac | interventions — Electrocardiography; Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cohort 1 (Other): This will include subjects with no known history of AF and are in normal sinus rhythm at time of screening
  Interventions: Device: 1-lead ECG
- Cohort 2 (Other): This will include subjects with known persistent or permanent AF who are in AF at the time of screening
  Interventions: Device: 1-lead ECG

INTERVENTIONS:
Device: 1-lead ECG — 1 lead ECG - All participants will record three single-lead ECGs at rest and three single-lead ECGs after exercise.
  Intervention Other: Exercise - All participants will undergo three trials of exercise.
  Other interventions: 12-lead ECG - All participants will simultaneously record 12-lead ECGs during rest and exercise sessions.
  Other Names: 12- lead ECG; Exercise

SUMMARY:
The purpose of the study is to evaluate the performance of ECG classification algorithms and their ability to classify heart rhythms into multiple categories of rhythms and heart rates

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all the following inclusion criteria to be enrolled:

  1. Able to read, understand, and provide written informed consent
  2. Willing and able to participate in the study procedures as described in the consent form
  3. Individuals who are 22 years of age and older at time of screening
  4. Able to communicate effectively with and follow instructions from the study staff
  5. Have a wrist circumference between 130 mm and 245 mm (Measured at "band center" on the preferred wrist).
  6. Subjects enrolled into Cohort 1 must have no known medical history of AF and in normal sinus rhythm at the time of screening.
  7. Subjects enrolled into Cohort 2 must have a known diagnosis of persistent or permanent AF and be in AF at the time of screening.

Exclusion Criteria:

* Subjects must meet none of the following criteria to be enrolled:

  1. Physical disability that precludes safe and adequate testing
  2. Physical or medical impairments that preclude exercise testing such as musculoskeletal back pain, arthritis, leg claudication, etc.
  3. Mental impairment as determined by the Investigator
  4. Pregnant women at the time of the screening visit.
  5. Subjects with any Medical History, Physical exam, vital sign or any other study procedure finding/assessment that in the opinion of the investigator could compromise subject safety during study participation or interfere with the study integrity and/or the accurate assessment of the study objectives. This includes patients with known untreated medical conditions that are considered clinically significant by the Investigator, such as but not limited to significant anemia, important electrolyte imbalance and untreated or uncontrolled thyroid disease. Physical exam limitations include but not limited to open wound(s) on the wrist and forearm where the subject will be wearing the watch.
  6. Any history of wrist surgery with scarring in the area of the sensor location on the wrist where the subject will be wearing the watch
  7. Vital signs measurement, medical history, or physical exam finding that makes the subject inappropriate for participation according to the Investigator.
  8. Tattoos or moles in the area of the sensor location on the wrist where the subject will be wearing the watch.
  9. Skin conditions on either wrist that would preclude subject from wearing watch on either wrist. Severe symptomatic (or active) overly dry/injured skin, skin disorders, or allergic skin reactions such as eczema, rosacea, impetigo, dermatomyositis or allergic contact dermatitis on wrist and locations where the electrodes will be placed (e.g. chest, forearms, stomach), as determined by the investigator.
  10. Known allergy or significant sensitivity to medical adhesives, isopropyl alcohol, or ECG patch
  11. Known allergy or sensitivity to fluorocarbon-based synthetic rubber, such as fluoroelastomer bands primarily used in the wrist worn fitness devices.
  12. Clinically significant hand tremors as judged by the Investigator.
  13. Participation in a previous study that involved a wrist-worn ECG device.
  14. Subjects with implanted cardiac devices such as a Pacemaker or an automated Implantable Cardioverter - Defibrillator

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Hope Research Institute, Phoenix, Arizona
  - Clinical Research of South Florida, Coral Gables, Florida
  - American Health Network of Indiana LLC, Avon, Indiana
  - Heartland Cardiology, Wichita, Kansas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: This will include subjects with no known history of AF and are in normal sinus rhythm at time of screening
  1-lead ECG: 1 lead ECG - All participants will record three single-lead ECGs at rest and three single-lead ECGs after exercise.
  Intervention Other: Exercise - All participants will undergo three trials of exercise.
  Other interventions: 12-lead ECG - All participants will simultaneously record 12-lead ECGs during rest and exercise sessions.
- Cohort 2: This will include subjects with known persistent or permanent AF who are in AF at the time of screening
  1-lead ECG: 1 lead ECG - All participants will record three single-lead ECGs at rest and three single-lead ECGs after exercise.
  Intervention Other: Exercise - All participants will undergo three trials of exercise.
  Other interventions: 12-lead ECG - All participants will simultaneously record 12-lead ECGs during rest and exercise sessions.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 241 | 305
Completed | 241 | 293
Not Completed | 0 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 241 | 305 | 546
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 207 | 80 | 287
  >=65 years | 34 | 225 | 259
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.1 (15.92) | 69.7 (9.35) | 58.0 (18.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 76 | 205
  Male | 112 | 229 | 341
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 99 | 71 | 170
  Ethnicity: Not Hispanic or Latino | 142 | 234 | 376
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 13 | 1 | 14
  Race: Black or African American | 35 | 4 | 39
  Race: Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Race: White | 185 | 298 | 483
  Race: More than one race | 2 | 1 | 3
  Race: Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 241 | 305 | 546

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Trials With Correct Classification of Normal Sinus Rhythm on Simultaneous 12-lead ECG as "Sinus Rhythm" or "High Heart Rate" on a Readable and Classifiable ECG App Strip.
Description: Specificity of sinus rhythm classification
Time Frame: 1 Day
Population: Subjects in each cohort include up to 2 trial measurements (at rest; after exercise). Overall number of units represents the number of trials rather than number of subjects.
Measure: Number; unit: percentage of trials
Units Other Than Participants: Trials
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 241 | 293
Number analyzed (Trials) | 429 | 10
percentage of trials | 99.3 | 100

2. Primary Outcome: Percentage of Trials With Correct Classification of AF on Simultaneous 12-lead ECG as "AF" on a Readable and Classifiable ECG App Strip.
Description: Sensitivity of sinus rhythm classification
Time Frame: 1 Day
Population: as for outcome 1
Measure: Number; unit: percentage of trials
Units Other Than Participants: Trials
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 241 | 293
Number analyzed (Trials) | 1 | 480
percentage of trials | 100 | 98.5

3. Secondary Outcome: Percentage of Trials With Correct Classification of Normal Sinus Rhythm at Normal Heart Rates as "Sinus Rhythm" on a Readable and Classifiable ECG App Strip
Time Frame: 1 Day
Population: as for outcome 1
Measure: Number; unit: percentage of trials
Units Other Than Participants: Trials
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 241 | 293
Number analyzed (Trials) | 228 | 6
percentage of trials | 98.2 | 100

4. Secondary Outcome: Percentage of Trials With Correct Classification of AF at Normal Heart Rates as "AF" on a Readable and Classifiable ECG App Strip
Time Frame: 1 Day
Population: as for outcome 1
Measure: Number; unit: percentage of trials
Units Other Than Participants: Trials
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 241 | 293
Number analyzed (Trials) | 1 | 274
percentage of trials | 100 | 98.9

5. Secondary Outcome: Percentage of Trials With Correct Classification of Sinus Tachycardia at High Heart Rates as "High Heart Rate" on a Readable and Classifiable ECG App Strip
Time Frame: 1 Day
Population: as for outcome 1
Measure: Number; unit: percentage of trials
Units Other Than Participants: Trials
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 241 | 293
Number analyzed (Trials) | 201 | 4
percentage of trials | 90.5 | 100

6. Secondary Outcome: Percentage of Trials With Correct Classification of AF at High Heart Rates as "AF (High Heart Rate)" on a Readable and Classifiable ECG App Strip
Time Frame: 1 Day
Population: as for outcome 1
Measure: Number; unit: percentage of trials
Units Other Than Participants: Trials
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 241 | 293
Number analyzed (Trials) | 0 | 206
percentage of trials |  | 83

7. Secondary Outcome: Percentage of Trials With Equivalence of the ECG App Waveform to Lead I From a 12-lead ECG as Measured by Acceptable Morphology of PQRST Complexes
Description: A "pass" rating is given when the waveforms of the ECG tracings generated by the algorithm and the Lead 1 of the 12-Lead ECG appear to overlay to the unaided eye. The morphology of the waveforms will be considered equivalent if at least 80% of the paired waveforms for the first 6 PQRST complexes are given a "pass" rating.
Time Frame: 1 Day
Measure: Number; unit: percentage of trials
Units Other Than Participants: Trials
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 45 | 48
Number analyzed (Trials) | 84 | 94
percentage of trials | 100 | 100

8. Secondary Outcome: Percentage of Trials With Equivalence of the ECG App Waveform to Lead I From a 12-lead ECG as Measured by R-Wave Amplitude Agreement
Description: A "pass" rating is given when the difference of the R-wave amplitudes (typically the highest peak of one cardiac rhythm cycle) between the ECG tracings generated by the algorithm and the Lead 1 of the 12-Lead ECG is <= 2mm. The R-wave amplitude agreement will be considered equivalent if at least 80% of the largest R-wave amplitudes of the paired waveforms are given a "pass" rating.
Time Frame: 1 Day
Population: as for outcome 1
Measure: Number; unit: percentage of trials
Units Other Than Participants: Trials
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 45 | 48
Number analyzed (Trials) | 84 | 94
percentage of trials | 96.4 | 97.9

ADVERSE EVENTS:
Time Frame: 1 Day
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/241 | 0/305
Serious Adverse Events (participants affected / at risk) | 0/241 | 0/305
Other Adverse Events (participants affected / at risk) | 1/241 | 0/305
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=241) | Cohort 2 (N=305)
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT04247581/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT04247581/SAP_001.pdf